CLINICAL TRIAL: NCT06982937
Title: A Mechanistic Perspective on Post-Activation Performance Enhancement Responsiveness: A Randomized Controlled Study of Acute Changes in Muscle Architecture, Contractile Property Kinetics, and Muscle Excitability
Brief Title: Mechanistic Drivers of Acute PAPE Responsiveness: Muscle Architecture, Contractile Kinetics, and Excitability in a Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Jerzy Kukuczka Academy of Physical Education in Katowice (Other)
Responsible Party: Principal Investigator, Artur Terbalyan, PhD student, lecturer, The Jerzy Kukuczka Academy of Physical Education in Katowice
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 01/2023
Record Dates: First submitted 2025-05-05; First posted 2025-05-21 (Actual); Results first posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-11

CONDITIONS: Neuromuscular Function; Muscle Activation; Postactivation Potentiation; Ultrasonography; Tensiomyography; Contraction; MHC-I
Keywords: MHC-I; Tensiomyography; Ulstrasonography; Electromyogpraphy; Postactivation potentiation; PAPE

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Half-Squat (Experimental): Participants perform one set half-squats using a free-weight barbell in a squat rack to elicit PAPE
  Interventions: Other: High-Intensity Half-Squat
- Treadmill running (Active Comparator): Participants jogged on a level treadmill for five minutes at a comfortable pace to provide general muscle warm-up without significant neuromuscular priming.
  Interventions: Other: Treadmill running

INTERVENTIONS:
Other: High-Intensity Half-Squat — Participants in the conditioning arm perform a single set of two to three half-squats with a free-weight barbell set at 90% of their one-rep max (1RM). Each squat is taken down until the thigh is parallel to the floor (knee at ~90°) and then driven upward as explosively as possible.
  Arms: High-Intensity Half-Squat
Other: Treadmill running — Participants engaged in a standardized 5-minute treadmill warm-up. Participants were instructed to walk at a moderate, self-selected pace of approximately 7-9 km/h, maintaining an incline of 0%. Heart rate and perceived exertion were monitored to ensure that the activity remained within a light-intensity range (Borg scale: 6-11).
  Arms: Treadmill running

SUMMARY:
The goal of this study is to find out if one short set of heavy half-squats can help football players jump higher right away-and to understand what happens inside their muscles and nerves to make that boost happen.

Key questions

* Will performing 2-3 half-squats at 90% of one-rep max give a bigger jump boost than jogging on a treadmill for five minutes?
* After each warm-up, how do muscle speed and stiffness, muscle size and fiber angle, and nerve signals change over the next 12 minutes?
* Does each player's contribution of fast and slow muscle fibers affect how much and how long their jump improves?

Study Plan Researches will invite 44 healthy football players, ages 18-21, who train regularly and meet our health rules. No one will know which warm-up each player does until the end.

Participants will:

* Get baseline tests of jump height, muscle speed and stiffness (using a harmless electrical sensor), muscle size and fiber angle (using ultrasound), and nerve signals (using sticky pads on the skin).
* Be randomly assigned to either:

  1. Heavy-squat group: 2-3 half-squats at 90% of their one-rep max
  2. Jogging group: easy jog or walk on a treadmill for five minutes
* Repeat all tests right after the warm-up and again at 4, 6, 8, 10, and 12 minutes to see how jump height and all muscle and nerve measures change over time.
* Have their muscle fiber mix estimated from the first muscle-speed test to see if fiber type explains who gets the biggest jump boost.

All tests are safe, painless, and approved by an ethics board. Players can stop at any time without giving a reason. This study will help athletes and coaches choose the best warm-up to get stronger, faster jumps right before a game or practice.

DETAILED DESCRIPTION:
Design and setting. The study will be a randomized, assessor-blinded, parallel-group trial conducted in university sport-science laboratories. Two arms will be used: a heavy half-squat conditioning activity and an active warm-up control. All procedures will follow written standard operating protocols.

Participants. Healthy, 44 resistance-trained male football/soccer players will be screened and will provide written informed consent. Eligibility will require regular training and the absence of musculoskeletal, neurological, dermatological, or cardiovascular contraindications to high-intensity exercise or peripheral electrical stimulation. Testing will be scheduled on a consistent team microcycle day to control for prior load.

Visit schedule. Visit 1 - Familiarization and strength assessment. Medical screening, anthropometrics, and a progressive half-squat session will determine individual one-repetition maximum (1RM). Squat depth will be standardized at approximately 90° knee flexion with rack pins and spotters.

Visit 2 - Experimental session. After compliance checks (sleep, diet, caffeine), participants will complete a structured general warm-up. Baseline tensiomyography (TMG) of the dominant vastus lateralis (VL), surface electromyography (EMG) normalization to maximal voluntary contraction (MVC), and baseline countermovement-jump (CMJ) testing will be completed. The allocated intervention will be delivered, followed by repeated CMJ testing with concurrent EMG at one-minute intervals. Ultrasound imaging will be obtained at baseline and after the final CMJ series.

Arms and interventions. Experimental arm (conditioning activity). One set of 2-3 free-weight half-squats at ~90% 1RM will be performed from a rack with spotter supervision.

Control arm (active warm-up). Approximately five minutes of treadmill running at light-moderate intensity (0% incline) will be completed.

Outcome measures and timing. Primary outcome. Change in CMJ height at each minute from 4 to 12 minutes after the intervention, relative to baseline (5 prespecified post-intervention time points at 2-min resolution).

CMJ-derived flight time, take-off velocity (device-derived where available), and individualized responder categorization at each minute using a predefined smallest-detectable-change threshold anchored to familiarization reliability.

Exploratory relationships between neuromuscular phenotype (TMG) and the magnitude/timing of CMJ responses.

Exploratory changes in VL architecture (ultrasound thickness, pennation, derived fascicle length) across the session.

Electromyography outcome (recorded for every jump). For every CMJ, surface EMG amplitude will be recorded and expressed as a percentage of the participant's maximal voluntary contraction (%MVC). The primary EMG variables will be RMS EMG (%MVC) across the propulsive phase and peak RMS (%MVC) within the final 200-250 ms before take-off.

Following the intervention, one CMJ will be performed at minute 1 and subsequently at each exact minute through minute 12. If a jump is technically invalid, a single replacement attempt will be permitted within that minute. Standardized instructions and hand placement will be maintained for all trials.

Instrumentation and standardization. CMJ. Jumps will be measured with a validated optical timing system on a non-slip surface. Foot placement and countermovement depth will be self-selected but replicated across trials.

Electromyography. Wireless surface EMG will be recorded from VL (with optional rectus femoris and biceps femoris for context). Skin will be shaved, lightly abraded, and cleaned with alcohol; disposable Ag/AgCl electrodes with ~20-mm inter-electrode distance will be placed along the fiber direction following SENIAM guidance and skin-marked for repeatability. Signals will be sampled at ≥2,000 Hz, band-pass filtered 20-450 Hz, notch-filtered at mains frequency, full-wave rectified, and converted to RMS with a 50-ms window. EMG and CMJ timing will be synchronized via hardware trigger; take-off will be identified from the optical system to define the propulsive phase. Prior to experimental jumps, three 3-5 s isometric knee-extension MVCs at ~60° knee flexion will be performed against a fixed dynamometer or rigid strap with strong verbal encouragement and 2-3 min rests. The highest stable 500-ms RMS epoch will define 100% MVC for normalization.

Tensiomyography. VL contractile properties (Td, Tc, Tr, Ts, Dm, and displacement-rate metrics) will be obtained with a displacement sensor at constant pre-tension. Participants will be supine with the knee supported at ~120°. Electrode positions will be standardized and skin-marked; single twitches will be delivered with inter-stimulus intervals ≥10 s. A validated multivariable model will estimate %MHC-I as a non-invasive phenotype proxy.

Ultrasound. B-mode imaging with a linear-array transducer will quantify VL thickness and pennation at mid-thigh; probe alignment will follow fascicle direction with minimal gel and consistent pressure. Fascicle length will be estimated from thickness and pennation. Three longitudinal images per site will be acquired and averaged.

Randomization and masking. Participants will be randomized using concealed, sequentially numbered envelopes prepared by personnel independent of data collection. CMJ/EMG assessors will be blinded to allocation and will operate in a separate space from the intervention station. Data files will contain coded identifiers only.

Participant flow during Visit 2. Participants will arrive for compliance checks. A standardized warm-up will be performed. MVC procedures for EMG normalization will be completed. Baseline TMG and baseline CMJ with EMG will be recorded. The allocated intervention will be administered. CMJ with EMG will be recorded at minutes 1-12. Ultrasound imaging will be performed at the end of the series, followed by cool-down and debrief.

Responder framework. At each minute, CMJ change will be classified for individual interpretation as positive, no-change, or negative using a priori smallest-detectable-change thresholds derived from familiarization reliability.

Safety and risk mitigation. Heavy squats will be performed in racks with pins and spotters; participants will have been familiarized with high loads during Visit 1. TMG will use brief single twitches with conservative current progression and long inter-stimulus intervals. Surface EMG and ultrasound are non-invasive; electrode preparation and probe handling will follow hygienic and standardized procedures. Adverse events and discomfort will be documented, and testing will cease if safety concerns arise.

Data capture and quality assurance. All devices will be calibrated before each session. Electrode and probe sites will be marked to ensure within-session consistency. Operators will complete training and inter-rater checks before data collection. Raw data will be stored on encrypted, access-controlled servers with audit trails. Predefined rules will govern artifact handling, trial acceptance, and protocol deviations.

Confidentiality and data handling. Participant identities will be coded. Source documents and electronic records will be stored on encrypted drives with restricted access limited to authorized personnel.

Discontinuation and withdrawal. Participants may withdraw at any time. Investigators will discontinue participation in the case of adverse signs, illness, or non-compliance. Data collected to the point of withdrawal will be retained unless the participant requests removal under the approved ethics framework.

ELIGIBILITY:
Inclusion Criteria:

* Male football players aged 18-23 years
* Minimum of 3 structured training sessions per week for the past 6 months
* No history of lower-limb musculoskeletal injuries (e.g., ligament sprain, muscle tear) within the past 2 months
* No diagnosed dermatological conditions affecting electrode placement (e.g., psoriasis, eczema)
* No cardiovascular disease (e.g., hypertension, arrhythmia)
* No neuromuscular disorders (e.g., neuropathy, myopathy) on clinical examination
* Able to complete a 1RM half-squat protocol and countermovement jump without pain

Exclusion Criteria:

* Use of performance-enhancing supplements/medications within 2 weeks prior to enrollment
* Missed more than 4 scheduled training sessions per month over the past 2 months
* Blood pressure >140/90 mmHg at rest or resting heart rate >90 bpm
* Any contraindication to electrical stimulation (e.g., pacemaker, implanted metal device)
* Failure to provide written informed consent or withdrawal of consent at any time

Ages: 18 Years to 23 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is restricted to participants who are biologically male and self-identify as male
Enrollment: 44 (Actual)
Dates: Start 2025-02-02 (Actual); Primary Completion 2025-06-25 (Actual); Study Completion 2025-07-25 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Jerzy Kukuczka Academy of Physical Education in Katowice, Katowice, Silesian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No
Data collected during this study will be available upon reasonable request. Individual participant data sharing will be considered on a case-by-case basis, subject to ethical approval, participant consent, and data protection regulations. Data requests must clearly outline the purpose, intended analyses, and measures taken to ensure confidentiality and data security.

REFERENCES:
- [Background] Simunic B, Degens H, Rittweger J, Narici M, Mekjavic IB, Pisot R. Noninvasive estimation of myosin heavy chain composition in human skeletal muscle. Med Sci Sports Exerc. 2011 Sep;43(9):1619-25. doi: 10.1249/MSS.0b013e31821522d0. PMID 21552151

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Intensity Half-Squat | Treadmill Running | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 22 | 44
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 22 | 22 | 44
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 22 | 22 | 44
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Poland | 22 | 22 | 44
%MHC-1 [Mean (Standard Deviation); unit: %] — Non-invasively estimated percentage of myosin heavy chain type I (MHC-I) isoform in the vastus lateralis muscle. The prediction is based on muscle characteristics obtained at rest during standardized TMG testing, using a previously developed regression model (Simunić, 2011).
  % | 26.14 (9.19) | 27.28 (10.01) | 26.71 (9.6)
Contraction time [Mean (Standard Deviation); unit: ms] — Contraction time of the vastus lateralis muscle, defined as the time interval between reaching 10% and 90% of peak radial muscle displacement following a single supramaximal electrical stimulus. The measure is obtained from the displacement-time curve recorded by a non-invasive muscle displacement sensor placed over the muscle belly during standardized TMG testing. Shorter contraction times are typically associated with a greater proportion of fast-twitch fibres, whereas longer contraction times reflect slower contractile properties.
  ms | 26.34 (2.15) | 23.01 (1.08) | 24.68 (0.76)
Delay time [Mean (Standard Deviation); unit: ms] — Delay time of the vastus lateralis muscle, defined as the time interval between the electrical stimulus and the moment when radial muscle displacement reaches 10% of its maximal value. The variable is derived from the same displacement-time curve as contraction time and reflects the electromechanical delay between stimulation and the onset of mechanical response.
  ms | 23.47 (1.16) | 21.91 (1.14) | 22.69 (0.02)
Muscle displacement [Mean (Standard Deviation); unit: mm] — Maximal radial muscle displacement of the vastus lateralis during a single supramaximal electrical stimulus/ Higher values indicate greater transverse deformability of the muscle-tendon unit, which is commonly interpreted as reflecting lower passive stiffness and/or lower muscle tone, whereas lower values suggest a stiffer muscle-tendon complex.
  mm | 6.78 (1.93) | 6.61 (1.59) | 6.70 (1.75)
Relaxation time [Mean (Standard Deviation); unit: ms] — Relaxation time of the vastus lateralis muscle, defined as the time interval from 90% to 50% of maximal radial displacement on the descending portion of the twitch response. This variable is calculated from the displacement-time curve and reflects the rate of muscle relaxation following peak contraction.
  ms | 18.25 (5.16) | 16.61 (3.82) | 17.44 (4.56)
Sustain time [Mean (Standard Deviation); unit: ms] — Sustain time of the vastus lateralis muscle, defined as the time interval during which radial muscle displacement is maintained between 50% of maximal displacement on the ascending limb and 50% of maximal displacement on the descending limb of the twitch curve. This measure describes how long the muscle maintains a substantial level of contraction during the mechanically induced twitch.
  ms | 40.37 (4.27) | 37.49 (4.13) | 38.94 (4.40)
Muscle thickness [Mean (Standard Deviation); unit: cm] | 2.47 (0.36) | 2.57 (0.28) | 2.53 (0.32)
Pennation angle [Mean (Standard Deviation); unit: degrees] — Pennation angle of the vastus lateralis muscle fibres, measured at rest using B-mode ultrasound imaging at a standardized site on the muscle belly. Pennation angle is defined as the angle between the muscle fascicles and the deep aponeurosis. Larger pennation angles are generally associated with greater physiological cross-sectional area and force-generating capacity.
  degrees | 13.76 (2.05) | 14.23 (1.75) | 14.00 (1.90)
Fascile lenght [Mean (Standard Deviation); unit: cm] — =MT/sin(PA)
  *MT - muscle thickness PA - pennation angle
  Fascicle length is defined as the length of a visible fascicle between the superficial and deep aponeuroses; when fascicles are not fully visible within the image, length is estimated by linear extrapolation following the fascicle trajectory. Longer fascicle lengths are typically associated with a greater muscle shortening velocity and range of motion.
  cm | 10.61 (2.02) | 10.67 (2.12) | 10.64 (2.04)
Maximal strength level [Mean (Standard Deviation); unit: kg] — Maximal strength level assessed under standardized half-squat testing with barbell
  kg | 98.07 (9.63) | 102.04 (16.14) | 100.06 (13.29)
Jump height [Mean (Standard Deviation); unit: cm] | 45.23 (4.95) | 47.52 (4.70) | 46.38 (4.91)
Muscle activation during countermovement jump [Mean (Standard Deviation); unit: percentage of MVC] — Surface electromyographic activity (voluntary activation level) of the vastus lateralis muscle recorded during a standardized countermovement jump. Higher values indicate greater muscle activation of the vastus lateralis during the jump, whereas lower values indicate reduced activation.
  Results presented as % from maximal voluntary contraction (MVC) during the procedure of normalization (locked at 90 degrees knee extension)
  percentage of MVC | 45.87 (12.78) | 44.16 (10.92) | 45.02 (11.78)

OUTCOME MEASURES:

1. Primary Outcome: Jump Height 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 45.34 (5.28) | 47.41 (5.13)

2. Primary Outcome: Jump Height 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 48.01 (5.13) | 47.41 (3.92)

3. Primary Outcome: Jump Height 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 47.08 (5.31) | 48.10 (4.60)

4. Primary Outcome: Jump Height 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 46.17 (5.17) | 47.59 (3.90)

5. Primary Outcome: Jump Height 12 Minute
Time Frame: 12 minute post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 45.27 (5.14) | 47.91 (4.27)

6. Primary Outcome: Muscle Thickness Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.95 (0.37) | 2.63 (0.33)

7. Primary Outcome: Muscle Thickness 4 Minute
Time Frame: 4 minute post-intervention (single session)
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.92 (0.35) | 2.58 (0.33)

8. Primary Outcome: Muscle Thickness 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.83 (0.37) | 2.58 (0.30)

9. Primary Outcome: Muscle Thickness 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.70 (0.36) | 2.53 (0.32)

10. Primary Outcome: Muscle Thickness 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.66 (0.35) | 2.60 (0.39)

11. Primary Outcome: Muscle Thickness 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 2.57 (0.44) | 2.55 (0.38)

12. Primary Outcome: Pennation Angle Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degrees | 17.83 (2.49) | 13.84 (1.98)

13. Primary Outcome: Pennation Angle 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: degress
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degress | 16.95 (2.63) | 13.37 (2.07)

14. Primary Outcome: Pennation Angle 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degrees | 17.09 (2.70) | 14.06 (2.39)

15. Primary Outcome: Pennation Angle 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degrees | 16.84 (2.88) | 14.09 (2.45)

16. Primary Outcome: Pennation Angle 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degrees | 16.52 (2.70) | 13.96 (2.42)

17. Primary Outcome: Pennation Angle 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
degrees | 14.61 (3.16) | 13.55 (2.62)

18. Primary Outcome: Fascicle Length Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 9.82 (1.88) | 11.26 (2.49)

19. Primary Outcome: Fascicle Length 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 10.27 (2.18) | 11.54 (3.17)

20. Primary Outcome: Fascicle Length 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 9.80 (1.64) | 10.86 (1.90)

21. Primary Outcome: Fascicle Length 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 9.59 (2.61) | 10.57 (1.60)

22. Primary Outcome: Fascicle Length 10 Minute
Time Frame: 10' minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 9.69 (2.46) | 10.97 (1.76)

23. Primary Outcome: Fascicle Length 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
cm | 10.69 (3.11) | 11.14 (1.98)

24. Primary Outcome: Muscle Activation During Countermovement Jump in 4 Minute
Description: Surface electromyographic activity (voluntary activation level) of the vastus lateralis muscle recorded during a standardized countermovement jump. Higher values indicate greater muscle activation of the vastus lateralis during the jump, whereas lower values indicate reduced activation.
  Results presented as % from maximal voluntary contraction (MVC) during the procedure of normalization (locked at 90 degrees knee extension)
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
percentage of MVC | 50.63 (14.18) | 43.96 (11.31)

25. Primary Outcome: Muscle Activation During Countermovement Jump in 6 Minute
Description: as for outcome 24
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
percentage of MVC | 45.29 (13.85) | 43.96 (11.31)

26. Primary Outcome: Muscle Activation During Countermovement Jump in 8 Minute
Description: as for outcome 24
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
percentage of MVC | 46.38 (13.61) | 49.43 (12.44)

27. Primary Outcome: Muscle Activation During Countermovement Jump in 10 Minute
Description: as for outcome 24
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
percentage of MVC | 48.76 (21.90) | 51.71 (14.85)

28. Primary Outcome: Muscle Activation During Countermovement Jump in 12 Minute
Description: as for outcome 24
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: percentage of MVC
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
percentage of MVC | 43.19 (9.49) | 34.39 (8.23)

29. Primary Outcome: Contraction Time Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 31.34 (2.94) | 29.04 (2.45)

30. Primary Outcome: Contraction Time 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 29.94 (2.61) | 27.91 (2.55)

31. Primary Outcome: Contraction Time 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 26.87 (2.32) | 27.98 (2.24)

32. Primary Outcome: Contraction Time 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 26.54 (2.33) | 26.43 (2.05)

33. Primary Outcome: Contraction Time 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 26.24 (2.35) | 26.83 (2.58)

34. Primary Outcome: Contraction Time 12 Minutes
Time Frame: 12 post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 26.01 (2.09) | 26.29 (1.77)

35. Primary Outcome: Delay Time Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 21.49 (1.16) | 22.54 (1.33)

36. Primary Outcome: Delay Time 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 21.06 (1.14) | 22.41 (1.35)

37. Primary Outcome: Delay Time 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 21.04 (1.18) | 22.52 (1.38)

38. Primary Outcome: Delay Time 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 20.77 (1.16) | 22.07 (1.36)

39. Primary Outcome: Delay Time 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 22.05 (2.39) | 22.84 (1.86)

40. Primary Outcome: Delay Time 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 21.70 (2.54) | 22.88 (1.91)

41. Primary Outcome: Relaxation Time Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 20.97 (7.46) | 16.35 (5.71)

42. Primary Outcome: Relaxation Time 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 19.08 (7.90) | 16.35 (5.71)

43. Primary Outcome: Relaxation Time 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 18.16 (7.52) | 17.57 (6.20)

44. Primary Outcome: Relaxation Time 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 19.28 (8.02) | 19.94 (8.53)

45. Primary Outcome: Relaxation Time 10 Minute
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 17.71 (7.14) | 16.63 (4.88)

46. Primary Outcome: Relaxation Time 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 17.20 (6.64) | 17.30 (5.48)

47. Primary Outcome: Muscle Displacement Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 5.70 (1.54) | 6.37 (1.35)

48. Primary Outcome: Muscle Displacement 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 5.98 (1.78) | 6.36 (1.46)

49. Primary Outcome: Muscle Displacement 6 Minute
Description: 6' post intervention measure
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 5.80 (1.19) | 6.83 (0.90)

50. Primary Outcome: Muscle Displacement 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 5.97 (1.34) | 6.59 (1.04)

51. Primary Outcome: Muscle Displacement 10 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 6.21 (1.43) | 6.22 (1.11)

52. Primary Outcome: Muscle Displacement 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
mm | 6.50 (1.55) | 6.23 (1.21)

53. Primary Outcome: Sustain Time Post
Time Frame: Immediate post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 48.86 (3.86) | 38.83 (2.77)

54. Primary Outcome: Sustain Time 4 Minute
Time Frame: 4 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 46.23 (3.74) | 39.52 (2.70)

55. Primary Outcome: Sustain Time 6 Minute
Time Frame: 6 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 43.27 (6.52) | 38.82 (4.52)

56. Primary Outcome: Sustain Time 8 Minute
Time Frame: 8 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 42.36 (4.33) | 39.03 (3.50)

57. Primary Outcome: Sustain Time 10 Minutes
Time Frame: 10 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 42.91 (5.47) | 39.11 (4.31)

58. Primary Outcome: Sustain Time 12 Minute
Time Frame: 12 minutes post-intervention
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | High-Intensity Half-Squat | Treadmill Running
Number analyzed (Participants) | 22 | 22
ms | 43.47 (4.97) | 40.77 (3.72)

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | High-Intensity Half-Squat | Treadmill Running
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
First, although outcome assessment was blinded, full double-blinding is pragmatically challenging in strength interventions and expectancy effects cannot be entirely excluded. Second, the fiber-type estimate pertains to a single muscle (VL), whereas CMJ performance reflects coordinated output from multiple muscle groups; generalizing VL composition to the whole task effector has inherent constraints. Finally, the MHC-I content of 26.14 ± 9.19% in the VL appears somewhat underestimated

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-18): https://cdn.clinicaltrials.gov/large-docs/37/NCT06982937/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/37/NCT06982937/ICF_001.pdf